CLINICAL TRIAL: NCT04537013
Title: A ProSpective, MulticEnter, Concurrently Controlled Clinical Study of Chondro-Gide® ArticUlar Cartilage CoveR for the Treatment of Large Chondral Lesions in the KnEe (SECURE)
Brief Title: Clinical Study of Chondro-Gide® for Large Chondral Lesions in the Knee
Acronym: SECURE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13575-237
Record Dates: First submitted 2020-08-18; First posted 2020-09-03 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-05

CONDITIONS: Knee Injuries; Cartilage Injury; Cartilage Disease; Knee Discomfort
Keywords: Microfracture; Cartilage; Knee
MeSH Terms: conditions — Knee Injuries; Cartilage Diseases; Fractures, Stress | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Control Arm (Active Comparator): Patients with small chondral lesions of the knee
  Interventions: Procedure: Microfracture
- Investigational Group (Experimental): Patients with large chondral lesions of the knee
  Interventions: Device: Microfracture plus placement of Chondro-Gide® ACC

INTERVENTIONS:
Procedure: Microfracture — Debridement of cartilage followed by placement of small holes in the effected area to fill the debrided area with marrow and cells.
  Arms: Control Arm
Device: Microfracture plus placement of Chondro-Gide® ACC — Debridement of cartilage followed by placement of small holes in the effected area to fill the debrided area with marrow and cells, followed by affixing Chondro-Gide® with fibrin glue.
  Arms: Investigational Group

SUMMARY:
Multi-center, prospective, concurrently controlled, non-randomized, double-blind (patient and assessor). Treatment of large chondral lesions in the knee with microfracture plus the Chondro-Gide® ACC is non-inferior to treatment of small chondral lesions treated with microfracture alone.

DETAILED DESCRIPTION:
The study evaluates the investigational treatment for treating large chondral lesions of the knee to the control treatment of microfracture alone for treating small lesions.Eligible patients with a large lesion will be treated with microfracture plus the Chondro-Gide® ACC and compared to patients with small lesions that are treated with microfracture alone. Outcome measures to be assessed include patient reported outcomes and freedom from certain adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. One symptomatic knee with cartilage defect on the medial femoral condyle, lateral femoral condyle, or trochlea, identified MRI or arthroscopy
3. Between 18 and 55 years of age
4. Subject is willing and able to comply with all study procedures, including visits, diagnostic procedures, and the rehabilitation protocol

Exclusion Criteria:

1. BMI ≥ 30 kg/m2
2. Symptomatic contralateral knee
3. Diagnosis of radiographic osteoarthritis with Kellgren-Lawrence grade 3 or more
4. Prior surgical treatment of the cartilage using microfracture, mosaicplasty, or autologous chondrocyte implantation (debridement and lavage are acceptable if the procedure was at least 3 months prior to enrollment)
5. Patella dysplasia
6. Chronic inflammatory arthritis or infectious arthritis
7. History of autoimmune disease or immunodeficiency
8. History of connective tissue disease
9. Intra-articular steroid use within the 3 months prior to enrollment
10. Other intra-articular injections (e.g. hyaluronic acid) within 3 months prior to enrollment
11. The patient is currently being treated with radiation, chemotherapy, immunosuppression or systemic steroid therapy with a dose equivalent to more than 5 mg prednisolone
12. Pregnancy or lack of adequate contraceptives if a female of child-bearing potential
13. Enrolled in another study, involved in the study (as a researcher/investigator/sponsor), or relative of someone directly involved in the study
14. Active infection of the index knee
15. Previous diagnosis of osteoporosis as diagnosed by DEXA, bone densitometry or CT scan
16. Any disorder or impairment that would interfere with evaluation of outcomes measures, such as neurological, degenerative muscular, psychiatric, or cognitive conditions
17. History or current substance or alcohol abuse as defined by the DSM-V
18. Any other medical condition that the investigator determines would interfere with the validity of the study
19. Known allergy to porcine collagen
20. Symptom duration greater than 36 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 234 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Patients achieving composite clinical success (CCS) at 24 months follow-up, with CCS | 24 Months
  The CCS is defined as a patient meeting all of the three following criteria:
  1. Improvement in the Pain sub-scale of the Knee Injury and Osteoarthritis Outcomes Score (KOOS) between baseline to 24 months follow-up
  2. Improvement in function, defined as an improvement in the International Knee Documentation Committee (IKDC) score between baseline to 24 months follow-up
  3. Freedom from device- or procedure-related serious adverse events (SAEs) or secondary surgical intervention related to the device, procedure, or treated lesion

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score | Baseline, 6 weeks, 3 months, 6 months, 12 months, 18 months, and 24 months
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a knee-specific instrument, developed to assess the patients' opinion about their knee and associated problems. The KOOS evaluates both short-term and long-term consequences of knee injury. Calculate the mean score of the individual items of each subscale and divide by 4 (the highest possible score for a single answer option). Traditionally in orthopedics, 100 indicates no problems and 0 indicates extreme problems.
Magnetic Resonance Observation of Cartilage Score | 3 months, 24 months
  Magnetic Resonance Image (MRI) will be obtain during the course of the study at 3 months and 24 months. MOCART 2.0 scoring will occur by independent assessment using the MOCART score. The score is a 9-part and 29-item scoring system, also resulting in a final cartilage repair tissue score between 0 and 100 points; 0 points represent the worst imaginable score, 100 points represent the best imaginable score.
Patient satisfaction | 6 weeks, 3 months, 6 months, 12 months, 18 months, and 24 months
  1. Were you satisfied with the procedure? (Satisfied, Somewhat satisfied, Neutral, Somewhat unsatisfied, Unsatisfied)
  2. Would you have this procedure again if needed on the other knee? (Definitely yes, Probably yes, Not Sure, Probably Not, Definitely Not)
Tegner Activity Scale | 6 weeks, 3 months, 6 months, 12 months, 18 months, and 24 months
  The Tegner activity score is a one-item score that grades activity based on work and sports activities. Tegner activity level scale is a scale that aims to provide a standardized method of grading work and sporting activities. A scale of the highest level activity being 10 and the lowest being 0
Employment status | Baseline, 6 weeks, 3 months, 6 months, 12 months, 18 months, and 24 months
  Employment status will be collected as: Employed full-time, Employed part-time, Not employed due to knee problems, Not employed due to reasons other than knee problems.
EuroQol-5 Dimension (EQ-5D) | Baseline, 6 weeks, 3 months, 6 months, 12 months, 18 months, and 24 months
  The EQ-5D measures as a descriptive system comprised of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: Fabiana Martinelli, Study Director — Geistlich Pharma AG; Kevin Plancher, MD, Principal Investigator — Plancher Orthopedics and Sports Medicine
Locations (15):
- United States (3):
  - The MORE Foundation, Phoenix, Arizona
  - Orthopaedic Foundation, Stamford, Connecticut
  - Emory Sports Medicine Complex, Johns Creek, Georgia
- Canada (6):
  - Fraser Orthopaedic Institute, New Westminster, British Columbia
  - University of Calgary, Calgary, CGY
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Sunnybrook Research Institute (SRI), Toronto, Ontario
  - University of Toronto Orthopaedics, Toronto, TOR
- Germany (6):
  - Gelenkzentrum Mittelrhein GmbH, Mayen, Mayen
  - Regio Kliniken GmbH, Pinneberg, Schleswig-Holstein
  - Universitätsklinikum Schleswig Holstein Campus Lübeck, Lübeck
  - Orthopädische Chirurgie München, München
  - Sportklinik Ravensburg, Ravensburg
  - University Hospital Regensburg, Regensburg

IPD SHARING:
Plan to Share IPD: No